CLINICAL TRIAL: NCT00129077
Title: Does the Use of a Moisture Chamber Decrease the Incidence of Corneal Abrasions in Critically Ill Pediatric Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Boston Children's Hospital (Other); Society of Critical Care Medicine (Other); American Association of Critical Care Nursing (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2003-12005
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-07

CONDITIONS: Eye Injuries; Critically Ill
Keywords: Pediatric critical care; neuromuscular blocking agents; corneal abrasions
MeSH Terms: conditions — Eye Injuries; Critical Illness; Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: plastic wrap over eye & lubrication applied q6 hrs

SUMMARY:
The purpose of this study is to identify the incidence of scratches on the surface of the eye in children who cannot blink due to medication use and to identify how best to reduce the risk of a scratch on the surface of the eye when patients are using specific medicines.

DETAILED DESCRIPTION:
Critically ill children may require neuromuscular blockade as a treatment modality. These children require careful eye care to prevent corneal abrasions. However, current evidence does not exist to guide best practices on eye care. This research study will evaluate 2 types of eye care therapy. The eyes will be randomly assigned to the control or experimental eye care therapy group. The control eye will receive lubricating ointment every 6 hours. The experimental eye will receive lubricating ointment every 6 hours and have a plastic covering to create a moisture chamber. Using daily fluorescein staining to detect corneal abrasions, each child will be studied for up to 9 days. Children who develop corneal abrasions will be discharged from the study and the primary care team will be notified. The two groups will then be compared to determine the therapy associated with the lowest incidence of corneal abrasions.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 42 weeks post-conceptual age and less than 18 years
* Anticipated need for neuromuscular blockade therapy for at least 24 hours

Exclusion Criteria:

* Use of continuous neuromuscular blockade therapy for more than 36 hours (early intervention study)
* Past medical history of abnormal blink reflex or incomplete lid closure
* History of daily eye drop use
* Facial trauma
* Alteration in periorbital skin integrity prohibiting eyelid closure or effective creation of a moisture chamber
* Known allergy to eye lubricant

Ages: 2 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2004-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Development of corneal abrasions | 9 days

SECONDARY OUTCOMES:
Incidence of corneal abrasions | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Martha AQ Curley, PhD, Study Chair — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts